CLINICAL TRIAL: NCT02864537
Title: Comparison Between Conventional Anticoagulation Treatment and Self-management of Anticoagulation Treatment
Brief Title: Self-management of Anticoagulation Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Una Ørvim Sølvik, Associate Professor, University of Bergen
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Lokkebo
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Atrial Fibrillation; Venous Thromboembolism; Artificial Heart Valve
Keywords: warfarin; self-management; Conventional management; Training; TTR; Complications; Quality of life
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional treatment (No Intervention): Conventional anticoagulation treatment Before enrolment
- Self-management (Experimental): Trained to monitor INR and dose warfarin
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — Patients were trained to measure INR and dose warfarin
  Arms: Self-management

SUMMARY:
The aim of the study was to compare self-management of anticoagulant treatment with conventional anticoagulant treatment in Norway.

DETAILED DESCRIPTION:
Patients (n=132) on anticoagulant treatment with warfarin participated in a 21 weeks training program where they learned how to analyse International Normalised Ratio (INR) using the point-of-care instrument CoaguChek®XS and dose warfarin. The patients had to display their skills through a test before considered self-managing. They continued to measure INR weekly for two years. All INR values during the training program and self-control period were collected. In addition, the patients were told to notify if they had any complications during this period. INR values and complications two years before enrolment was collected from INR cards and/or their general practioner. The participant filled in a quality of life-questioner at enrolment and after two years of self-management.

ELIGIBILITY:
Inclusion Criteria:

* On life-long oral anticoagulation therapy
* Judged to be qualified for patient self-management anticoagulation treatment by their GP
* Motivated to follow the training program

Exclusion Criteria:

* Drug abuse
* Liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in Time in therapeutic range (TTR) | From two years before enrolment until two years of self management
  Change in TTR from conventional treatment to self-management

SECONDARY OUTCOMES:
Change in number of complications | From two years before enrolment until two years of self management
  Compare number of complications during conventional treatment and during self-management
Quality of life (QoL) | Baseline before training and after two years with self-management

CONTACTS AND LOCATIONS:
Overall Officials: Una Ø Sølvik, PhD, Principal Investigator — University of Bergen

IPD SHARING:
Plan to Share IPD: Undecided